CLINICAL TRIAL: NCT06524947
Title: Phase III Clinical Trial to Evaluate the Protective Efficacy, Immunogenicity, and Safety of Quadrivalent Recombinant Norovirus Vaccine (Pichia Pastoris) Implanted in People Aged 6 Weeks to 13 Years
Brief Title: Clinical Trial of Protective Efficacy of Quadrivalent Recombinant Norovirus Vaccine (Pichia Pastoris)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LKM-2023-NoV01
Record Dates: First submitted 2024-07-19; First posted 2024-07-29 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Acute Gastroenteropathy Due to Norovirus
Keywords: prevention

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Infant experimental group (6 weeks -23 months) (Experimental): At least 6 weeks old but less than 2 years old.
  Interventions: Biological: quadrivalent recombinant norovirus vaccine (Pichia pastoris)
- Infant placebo control group (6 weeks -23 months) (Placebo Comparator): At least 6 weeks old but less than 2 years old.
  Interventions: Biological: quadrivalent recombinant norovirus vaccine (Pichia pastoris) placebo
- Toddler experimental group (2-5 years old) (Experimental): At least 2 years old but less than 6 years old.
  Interventions: Biological: quadrivalent recombinant norovirus vaccine (Pichia pastoris)
- Toddler placebo control group (2-5 years old) (Placebo Comparator): At least 2 years old but less than 6 years old.
  Interventions: Biological: quadrivalent recombinant norovirus vaccine (Pichia pastoris) placebo
- Children experimental group (6-13 years old) (Experimental): At least 6 years of age but under 14 years of age.
  Interventions: Biological: quadrivalent recombinant norovirus vaccine (Pichia pastoris)
- Children placebo control group (6-13 years old) (Placebo Comparator): At least 6 years of age but under 14 years of age.
  Interventions: Biological: quadrivalent recombinant norovirus vaccine (Pichia pastoris) placebo

INTERVENTIONS:
Biological: quadrivalent recombinant norovirus vaccine (Pichia pastoris) — Subjects were given three doses of quadrivalent recombinant norovirus vaccine (Pichia pastoris) at a 30-day interval.
  Main ingredients: recombinant ReNoV GI.1-VP1 protein, recombinant ReNoV GII.3-VP1 protein, recombinant ReNoVGII.4-VP1 protein, recombinant ReNoV GII.17-VP1 protein, aluminum hydroxide adjuvant, histidine, sodium chloride, tween 80, disodium phosphate, disodium hydrogen phosphate
  Arms: Children experimental group (6-13 years old); Infant experimental group (6 weeks -23 months); Toddler experimental group (2-5 years old)
Biological: quadrivalent recombinant norovirus vaccine (Pichia pastoris) placebo — Subjects were given three doses of quadrivalent recombinant norovirus vaccine (Pichia pastoris) placebo at a 30-day interval.
  Main ingredients: aluminum hydroxide adjuvant, histidine, sodium chloride, tween 80, disodium phosphate, disodium hydrogen phosphate
  Arms: Children placebo control group (6-13 years old); Infant placebo control group (6 weeks -23 months); Toddler placebo control group (2-5 years old)

SUMMARY:
The purpose of the research is to evaluate the protective efficacy, immunogenicity, and safety of quadrivalent recombinant norovirus vaccine (Pichia Pastoris) in people aged 6 weeks to 13 years.A total of 6600 infants and children aged 6 weeks to 13 years old were enrolled in this study, which were divided into 3 age groups: 1400 children (6-13 years old), 2200 toddler (2-5 years old), and 3000 infants (6-23 months old).Subjects of all ages were randomly assigned to the test group and the control group in a 1:1 ratio.All subjects received 3 doses of the experimental vaccine at 30 day intervals.

DETAILED DESCRIPTION:
Overall design: A multicenter, randomized, double-blind, placebo-controlled trial was designed.

The purpose of the research is to evaluate the protective efficacy, immunogenicity, and safety of quadrivalent recombinant norovirus vaccine (Pichia Pastoris) in people aged 6 weeks to 13 years.A total of 6600 infants and children aged 6 weeks to 13 years old were enrolled in this study, which were divided into 3 age groups: 1400 children (6-13 years old), 2200 toddler (2-5 years old), and 3000 infants (6-23 months old).Subjects of all ages were randomly assigned to the test group and the control group in a 1:1 ratio.All subjects received 3 doses of the experimental vaccine at 30 day intervals.

Protective effectiveness evaluation:All subjects entered the observation period 7 days after completing the first dose of immunization. Stool and/or vomit samples (if applicable) from all AGE cases occurring during the observation period were collected and AGE caused by Norovirus was identified by PCR.Primary protective efficacy was calculated using data from primary endpoint cases that occurred between 7 days after completion of full immunization and the end of the observation period.

Immunogenicity evaluation:For the immunogenic subgroup of subjects (120 subjects before the study number of each age group in a clinical trial site, a total of 360 subjects), blood samples were collected before the first dose of immunization, 31 days after the second dose of immunization, 31 days, 180 days, 1 year and 2 years after the total immunization, and blood samples were 2.5~3.0ml each time.It is used to detect anti-norovirus IgG antibody, tissue Blood group antigen (HBGA) blocking antibody, and to detect the immunogenicity of anti-norovirus.

Safety evaluation:Adverse events (AE) and serious adverse events (SAE) : All enrolled subjects collected AE 30 minutes after each dose of vaccine, enlisted AE 0-7 days, non-enlisted AE 0-30 days, and SAE from the first dose to 180 days after full immunization.

ELIGIBILITY:
Inclusion Criteria:

* 1.The subject's legal guardian agrees to participate in the trial (consent is also required for subjects 8 years of age and older), and can provide proof of legal identity, is fully informed and has signed an informed consent form, and understands and complies with the requirements of the trial protocol to participate in the follow-up visits.
* 2.The age of the subjects on the day of enrollment is not less than 6 weeks old and not more than 13 years old, regardless of gender.
* 3.Those younger than 12 months of age: 2.5kg ≤ birth weight ≤ 4.5kg, 37 weeks ≤ weeks of gestation ≤ 42 weeks, born in normal labor (excluding severe abnormal labor and history of severe asphyxia resuscitation).

Exclusion Criteria:

* 1.Allergic to or having a history of specific reactions to any component of the investigational vaccine; Previous history of severe allergy to any vaccine or drug (such as anaphylactic shock, laryngeal edema, anaphylactic purpura, local anaphylactic necrosis reaction (Arthus reaction), dyspnea, angioneurotic edema, etc.); People with allergic constitution.
* 2.A history of confirmed norovirus infection within 2 years.
* 3.Have a history of any of the following diseases or are suffering from serious diseases: ① Abnormal coagulation function: such as leukemia, congenital or acquired coagulation factor deficiency, aplastic anemia, thrombocytopenia and receiving anticoagulation therapy; ② Diseases affecting local observation: such as rational jaundice; ③Diseases affecting immune function: a history of congenital or acquired immunodeficiency or autoimmune disease; Uncontrolled lymphoproliferative diseases (such as chronic lymphocytic leukemia, Hodgkin's lymphoma, etc.); No spleen, or splenic surgery history, trauma history; ④Now suffering from infectious diseases: such as tuberculosis, viral hepatitis, etc； ⑤Neurological and psychiatric diseases: epilepsy, congenital brain hypoplasia, brain trauma, brain tumor, infection, brain nerve tissue damage caused by chemical and physical factors, etc., psychiatric history and family history； ⑥Other serious diseases that may interfere with the conduct or completion of the study: severe congenital malformations, severe developmental disorders, severe malnutrition, malignant tumors, congenital cardiovascular, liver, kidney diseases, etc.
* 4.Received blood or blood-related products (other than hepatitis B immunoglobulin) within 1 month prior to enrollment; Long-term use of systemic immunosuppressants or other immunomodulatory drugs within 3 months (defined as use for more than 14 days).
* 5.Have participated or are participating in other clinical trials (including drugs, biologics, or devices) within 3 months prior to enrollment.
* 6.The investigator believes that the subject has any disease or condition that could put the subject at risk, poor adherence or inability to complete the trial as required by the protocol, and conditions that interfere with the evaluation of vaccine response.

Ages: 6 Weeks to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6600 (Actual)
Dates: Start 2024-07-27 (Actual); Primary Completion 2027-03-28 (Estimated); Study Completion 2027-03-28 (Estimated)

PRIMARY OUTCOMES:
Protective efficacy against AGE caused by four genotypes of norovirus | From 7 days after full immunization to 2 years after 7 days after after full immunization
  Protective efficacy against AGE caused by the four genotypes included in the prophylactic vaccine (GI.1, GII.3, GII.4, GII.17) (co-infections of rotavirus and adenovirus were excluded) after 7 days of full immunization until the end of the observation period.Protective efficacy = 1 - (person-years of incidence in the vaccine group/person-years of incidence in the placebo group) × 100%; person-years of incidence = (number of cases of AGE (excluding co-infections with rotavirus and adenovirus) caused by the four genotypes included in the vaccine (GI.1, GII.3, GII.4, and GII.17) after 7 days of 3 doses of the vaccine/number of person-years of observation) × 100%.
Geometric mean titers (GMT) of IgG antibody | 31 days after 2 doses, 31 days after full immunization, 180 days after full immunization, 1 year, and 2 years after full immunization
  Geometric mean titers of IgG antibodies against norovirus (GI.1, GII.3, GII.4, GII.17) were measured at 31 days after 2 doses, 31 days after full immunization, 180 days after full immunization, 1 year, and 2 years after full immunization.
Geometric mean titers (GMT) of HBGA blocking antibody | at 31 days after 2 doses of immunization, 31 days after full immunization, 180 days after full immunization, 1 year, and 2 years after full immunization
  Geometric mean titers of HBGA blocking antibodies against norovirus (GI.1, GII.3, GII.4, GII.17) were measured at 31 days after 2 doses of immunization, 31 days after full immunization, 180 days after full immunization, 1 year, and 2 years after full immunization.
Positive conversion rate of IgG antibodies | 31 days after 2 doses, 31 days after full immunization, 180 days after full immunization, 1 year and 2 years after full immunization
  Positive conversion rate of IgG antibody against norovirus (GI.1, GII.3, GII.4, GII.17) at 31 days after 2 doses, 31 days after full immunization, 180 days after full immunization, 1 year and 2 years after full immunization.
Positive conversion rate of HBGA blocking antibody | 31 days after 2 doses of immunization, 31 days after full immunization, 180 days after full immunization, 1 year, and 2 years after full immunization
  The positive conversion rate of HBGA blocking antibodies against norovirus (GI.1, GII.3, GII.4, GII.17) was measured at 31 days after 2 doses of immunization, 31 days after full immunization, 180 days after full immunization, 1 year, and 2 years after full immunization.
Geometric mean titers Growth multiplier of IgG antibody | at 31 days after 2 doses of immunization and at 31 days after full immunization
  Geometric mean titers Growth multiplier of IgG antibody at 31 days after 2 doses of immunization and at 31 days after full immunization.
Geometric mean titers Growth multiplier of HBGA blocking antibody | at 31 days after 2 doses of immunization and at 31 days after full immunization
  Geometric mean titers Growth multiplier of HBGA blocking antibody at 31 days after 2 doses of immunization and at 31 days after full immunization.
Occurrence of any adverse event | within 30 minutes of each dose of vaccination
  Occurrence of any adverse event within 30 minutes of each dose of vaccination.
Occurrence of recruited adverse event | between day 0 and day 7 after each dose of vaccination
  Occurrence of recruited adverse event between day 0 and day 7 after each dose of vaccination.
Occurrence of non-recruited adverse event | between day 0 and day 30 after each dose of vaccination
  Occurrence of non-recruited adverse event between day 0 and day 30 after each dose of vaccination.
Occurrence of serious adverse event | from the first dose to 180 days after full immunization
  Occurrence of serious adverse event from the first dose to 180 days after full immunization.

CONTACTS AND LOCATIONS:
Overall Officials: teng huang, master, Principal Investigator — Guangxi Zhuang Autonomous Region Center for Disease Control and Prevention
Locations (3):
- China (3):
  - Guangxi Zhuang Autonomous Region Center for Disease Control and Prevention, Nanning, Guangxi
  - Hunan Center for Disease Control and Prevention, Changsha, Hunan
  - Sichuan Center for Disease Control and Prevention, Chengdu, Sichuan